CLINICAL TRIAL: NCT04931004
Title: Effect of Oral Hygiene Products on Reducing Expelled/Exhaled SARS-CoV-2
Brief Title: Oral Rinse to Reduced Expelled Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) During COVID-19 Infection
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Colgate Palmolive (Industry); University of Leicester (Other)
Responsible Party: Principal Investigator, Yingda L Xie, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Pro2020003236
Record Dates: First submitted 2021-06-16; First posted 2021-06-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Masking Description: Face mask and saliva SARS-CoV-2 viral RNA loads are measured before and after water rinse and before and after mouthwash rinse (intervention). Order is randomized. Participant is not told which rinse they are using, though can likely differentiate by taste.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 0.075% Cetylpyridinium Chloride (Experimental): Crossover design where a series of viral load measurements are taken before and after water rinse (placebo) and repeated before and after CPC rinse (intervention). The order of the rinses were randomized after the 19th participant.
  Interventions: Drug: Mouthwash Product

INTERVENTIONS:
Drug: Mouthwash Product — Commercially over-the-counter Colgate mouthwashes will be administered according to standard package instructions. Viral load will be measured prior to and after mouth rinse using serial face mask and saliva samples. Additionally viral load measured prior to and after water rinse using serial face mask and saliva samples. These serial measurements and both CPC and water rinses were conducted consecutively in one visit.
  Other Names: water rinse

SUMMARY:
Prospective, cross-sectional study evaluating the effect of commercially available mouthwashes on expelled/exhaled SARS-CoV-2 viral load using face mask sampling.

DETAILED DESCRIPTION:
The study will consist of a Control Phase to optimize procedures for measuring expelled/exhaled viral load, and a Evaluation phase comparing different commercially available mouthwashes.

In the Control Phase. up to 20 COVID-19 patients will be asked to undergo a sequence of face mask sampling and saliva collections prior to and after an oral rinse with (i) water and (ii) a commercially-available cetylpyridinium chloride (CPC) mouthwash.

Based on outcomes of the Control Phase, the study will proceed into the Evaluation Phase, which will randomize approximately 40 COVID-19 patients to receive 1 of 4 commercially available Colgate mouthwashes following standard package instructions. Face mask sampling and saliva will be collected prior to and after the mouth rinse to assess impact on SARS-CoV-2 viral load.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Able to provide consent
3. Polymerase chain reaction (PCR)-confirmed SARS-CoV-2 within previous 48 hours.

Exclusion Criteria:

1. Clinical contraindication or poor feasibility to complete study procedures
2. Unwilling or unable to produce saliva or face mask samples
3. Unable to produce at least 500 microliters of saliva.
4. Eaten within past 30 minutes
5. Known allergy to mouthwash products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Control Phase - Primary Endpoint | Single timepoint, ~1 hour
  Reduction in viral load by face mask sampling from pre-intervention to 0-15 with CPC versus water rinse control
Evaluation Phase - Primary Endpoint | Single timepoint, ~1.5 hours
  Reduction in viral load by face mask sampling from pre-intervention to 45-60 minutes versus water rinse control

SECONDARY OUTCOMES:
Evaluation Phase - Secondary Endpoint | Single timepoint, ~1 hour
  Reduction in viral load by face mask sampling from pre-intervention to 0-15 and15-30 minutes of oral rinse products versus water rinse control
Comparative Saliva Reduction | Single timepoint, ~1.5 hours
  Reduction in viral load in saliva pre-intervention to 30 and 60 minutes post-intervention.

OTHER OUTCOMES:
Influence of Speaking | Single timepoint, ~1 hour
  Difference in viral load by face mask sampling with speaking versus not speaking

CONTACTS AND LOCATIONS:
Overall Officials: Yingda L Xie, MD, Principal Investigator — Rutgers University; David Alland, MD, Principal Investigator — Rutgers University; Padmapriya Banada, PhD, Principal Investigator — Rutgers University
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal

DOCUMENTS (1):
  • Informed Consent Form (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT04931004/ICF_000.pdf